CLINICAL TRIAL: NCT03585361
Title: Utilizing All Health System Contacts to Offer Postpartum Family Planning (PPFP) to Pregnant Women and Women Within Twelve Months Postpartum in Ethiopia
Brief Title: Utilizing All Health System Contacts to Offer Postpartum Family Planning (PPFP) in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00007143
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Contraceptive Usage; Postpartum Family Planning; Contraception; Prenatal Care; Pregnancy
Keywords: Contraceptive Usage; Pregnancy; Postpartum Family Planning; Contraception; Prenatal Care; Postnatal Care; Postpartum Care; Family Planning; Ethiopia; Community Health Workers; Community Based Care; Health Extension Workers
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Health centers provide PPFP counseling and services, implementing current Government of Ethiopia policy and standard of care (including still experimental screening and intra-facility referrals of women bringing infants for immunization). Also, health centers conduct data reviews of PPFP counseling, intra-facility referrals and uptake data. At community level, HEWs provide PPFP counseling and services throughout continuum of care, volunteers (Development Army) promote PPFP, and HEWs and volunteers track PPFP method choice and uptake.
  Interventions: Behavioral: Health centers provide PPFP counseling and services; Behavioral: HEWs provide PPFP counseling and services; Behavioral: Volunteers (Development Army) promote PPFP; Behavioral: Health centers conduct data reviews; Behavioral: HEWs and volunteers track PPFP
- Comparison (Active Comparator): Health centers provide PPFP counseling and services, implementing current Government of Ethiopia policy and standard of care (including still experimental screening and intra-facility referrals of women bringing infants for immunization). Health centers conduct data reviews.
  Interventions: Behavioral: Health centers provide PPFP counseling and services; Behavioral: Health centers conduct data reviews

INTERVENTIONS:
Behavioral: Health centers provide PPFP counseling and services — Providers trained on PPFP counseling skills and insertion technique for placing intrauterine devices (IUDs) immediately after birth with a refresher on insertion techniques for IUDs and implants. Training also included how to use tools to document PPFP services and referrals. Follow up supervision ensured skill mastery and retention.
Behavioral: HEWs provide PPFP counseling and services — HEWs trained in PPFP counseling with a refresher on implant insertion skills. Training also included how to use tools to document PPFP services, method choice, and pregnancy risk at every contact during pregnancy and up to 12 months after birth. Follow up supervision ensured skill improvement and retention.
  Arms: Intervention
Behavioral: Volunteers (Development Army) promote PPFP — HEWs orient volunteers on promoting PPFP and how to use a pictoral tool to remind women to access ANC, immunization, and PPFP services and to document women's method preferences and pregnancy risk at every contact during pregnancy and up to 12 months after birth.
  Arms: Intervention
Behavioral: Health centers conduct data reviews — Health center staff document PPFP counseling, provision, and referrals in registers and use a facility dashboard to display and track aggregate PPFP data.
Behavioral: HEWs and volunteers track PPFP — HEWs and volunteers track PPFP counseling, choice of method, receipt of methods, and pregnancy risk starting in pregnancy through 12 months postpartum. HEWs and volunteers meet and review data.
  Arms: Intervention

SUMMARY:
This study is investigating whether use of postpartum family planning (PPFP) increases if messages on PPFP and, if desired, PPFP services are integrated into as many contacts as possible between women/couples and the health system during pregnancy and the first year after birth. Health system contacts may be at health facilities (including antenatal, labor and delivery, postnatal, and child immunization visits) or, with Ethiopia's Health Extension Program, at households or health posts in the community.

DETAILED DESCRIPTION:
This implementation research study used a quasi-experimental, mixed method design with two arms. Two districts in Arsi Zone in Ethiopia's Oromia Region (Hitosa and Lode Hitosa) were selected for the study. In each district, one primary health care unit (PHCU) - a public health center and its satellite health posts - was randomly assigned to the intervention arm and one to the comparison arm.

PPFP counseling, services, and documentation were strengthened through training and supervision at health centers in both intervention and comparison PHCUs, consistent with Government of Ethiopia policies and guidelines. Only the intervention arm received the community-based intervention. The community-based intervention involved training Health Extension Workers (HEWs) who staff health posts, make outreach home visits, and support volunteers under the government's Development Army. HEWs were trained on PPFP with a refresher on implant insertion. The community invention also involved giving tools to HEWs and volunteers to help them track women's PPFP preferences and pregnancy risk.

The study objectives are to:

1. Assess the effect of systematically integrating PPFP messages into contacts with the health system on uptake of PPFP through 12 months postpartum using a 'dose-response' analysis based on the number of contacts
2. Estimate the added effect of the community-based intervention by comparing uptake of PPFP through 12 months postpartum in intervention and comparison sites
3. Explore the acceptability and feasibility of tracking PPFP and reviewing data at health centers and HEWs and volunteers using record keeping and review processes to track women's decision-making and contraceptive use from pregnancy through 12 months postpartum
4. Explore factors influencing women's/couples' adoption of PPFP during the first 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. Women

   * Pregnant at time of enrollment
   * Willing to give informed consent
2. Provider interviews

   * Providers providing PPFP messages or services in study area
   * Willing to give informed consent

Exclusion Criteria:

1. Women

   * Not pregnant at time of enrollment
   * Living outside study area
2. Provider interviews

   * Not working in antenatal, labor & delivery, postnatal, or immunization care

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
PPFP uptake | 12 months after birth
  Proportion of interviewed postpartum women who used a modern family planning method within 12 months after giving birth

SECONDARY OUTCOMES:
Method choice | 12 months after birth
  Proportion of interviewed postpartum women who chose a method prior to delivery

CONTACTS AND LOCATIONS:
Locations (6):
- Ethiopia (6):
  - Boru PHCU, Hitosa, Oromiya
  - Sibu PHCU, Hitosa, Oromiya
  - Aleko PHCU, Lode Hitosa, Oromiya
  - Huruta PHCU, Lode Hitosa, Oromiya
  - Ligaba PHCU, Lode Hitosa, Oromiya
  - Lode Jimata, Lode Hitosa, Oromiya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pfitzer A, Jima GH, Sitrin D, Ayalew F, Ahmed S. Effect of multiple counselling contacts along the continuum of care on use of postpartum family planning in a cohort of Ethiopian women: a dose-response analysis. BMJ Open. 2024 Dec 20;14(12):e084247. doi: 10.1136/bmjopen-2024-084247. PMID 39806635

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT03585361/SAP_001.pdf
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT03585361/Prot_002.pdf